CLINICAL TRIAL: NCT05289661
Title: Descemet Endothelial Thickness Comparison Trials (DETECT I & II)
Brief Title: Descemet Endothelial Thickness Comparison Trial I
Acronym: DETECT I
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Oregon Health and Science University (Other); University of California, San Francisco (Other); University of California, Davis (Other); Case Western Reserve University (Other); Dartmouth-Hitchcock Medical Center (Other); University of Pennsylvania (Other); University of Miami (Other); Wills Eye Hospital (Unknown)
Responsible Party: Principal Investigator, Jennifer Rose-Nussbaumer, Associate Professor, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220590-I
Record Dates: First submitted 2022-03-02; First posted 2022-03-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Fuchs
MeSH Terms: interventions — K-115

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- UT-DSAEK plus topical ripasudil (Experimental): This arm will receive UT-DSAEK plus topical ripasudil 0.4%
  Interventions: Drug: Topical Ripasudil
- UT-DSAEK plus topical placebo (Placebo Comparator): This arm will receive UT-DSAEK plus topical placebo
  Interventions: Drug: Topical Placebo
- DMEK plus topical ripasudil (Experimental): This arm will receive DMEK plus topical ripasudil 0.4%
  Interventions: Drug: Topical Ripasudil
- DMEK plus topical placebo (Placebo Comparator): This arm will receive DMEK plus topical placebo
  Interventions: Drug: Topical Placebo

INTERVENTIONS:
Drug: Topical Ripasudil — To determine the effect of rho-kinase inhibitors on endothelial cell loss
  Other Names: Ripasudil
  Arms: DMEK plus topical ripasudil; UT-DSAEK plus topical ripasudil
Drug: Topical Placebo — topical Placebo
  Other Names: Placebo
  Arms: DMEK plus topical placebo; UT-DSAEK plus topical placebo

SUMMARY:
Descemet Endothelial Thickness Comparison Trial (DETECT) I is a multi-center, outcome assessor-masked, placebo-controlled clinical trial randomizing 160 patients in a 2x2 factorial design. The purpose of this study is to determine differences in visual outcomes between two types of corneal transplant surgeries, ultrathin Descemet stripping automated endothelial keratoplasty (UT-DSAEK) and Descemet membrane endothelial keratoplasty (DMEK), and to determine the effect of rho-kinase inhibitors on endothelial cell loss.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional endothelium from Fuchs Endothelial Corneal Dystrophy (FECD) with guttata extending beyond 4.5 mm of the central cornea or severe edema without visualization of guttata
* Dysfunctional endothelium from Pseudophakic Corneal Edema (PCE) or Iridocorneal Endothelial Syndrome (ICE) or other primary endothelial dysfunction such as Posterior Polymorphous Corneal Dystrophy (PPMD)
* Dysfunctional endothelium from prior graft failure after PKP or EK
* Controlled uveitis (defined as quiet for > 3 months off of topical steroids with or without systemic immunosuppression) or no uveitis
* Controlled glaucoma with topical medications and/or prior trabeculectomy or tube shunt without ongoing hypotony (IOP < 5 mmHg) or no glaucoma
* Good candidate for corneal transplantation for either DMEK or UT-DSAEK
* Willingness to participate
* Age greater than 18 years

Exclusion Criteria:

* Aphakia, or anterior chamber IOL or scleral fixated IOL in study eye prior to or anticipated during EK
* Pre-operative central sub-epithelial or stromal scarring that the investigator believes is visually significant and could impact post-operative stromal clarity assessment
* Peripheral anterior synechiae (iris to angle) in the angle greater than a total of three clock hours
* Visually significant optic nerve (ok to have small visual field defects) or macular severe pathology
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Best spectacle-corrected visual acuity (BSCVA) | 12 months
  Best spectacle-corrected visual acuity
Endothelial cell loss | 12 months
  Change between endothelial density at baseline versus density at 12 months

SECONDARY OUTCOMES:
Best spectacle-corrected visual acuity (BSCVA) | 3, 6 and 24 months
  Best spectacle-corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Stanford University, Palo Alto, California
  - University of California Davis, Sacramento, California
  - University of Miami, Palm Beach Gardens, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania